CLINICAL TRIAL: NCT06105983
Title: A PHASE 1, OPEN-LABEL, TWO-PERIOD, FIXED SEQUENCE STUDY TO INVESTIGATE THE EFFECT OF A PROTON PUMP INHIBITOR ON THE PHARMACOKINETICS OF SISUNATOVIR IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How a Medicine That Reduces Stomach Acid Affects the Level of Sisunatovir in the Blood of Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C5241017; 2023-507116-12-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — sisunatovir; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A (Experimental): Part 1: Sisunatovir without rabeprazole
  Interventions: Drug: Sisunatovir
- Treatment B (Active Comparator): Part 1: Sisunatovir with 40 mg rabeprazole
  Interventions: Drug: Sisunatovir; Drug: Rabeprazole 40 mg
- Treatment C (Active Comparator): Part 2: Sisunatovir suspension without rabeprazole
  Interventions: Drug: Sisunatovir suspension
- Treatment D (Experimental): Part 2: Sisunatovir suspension with 20 mg rabeprazole
  Interventions: Drug: Sisunatovir suspension; Drug: Rabeprazole 20 mg
- Treatment E (Experimental): Part 2: Sisunatovir suspension with 40 mg rabeprazole
  Interventions: Drug: Rabeprazole 40 mg; Drug: Sisunatovir suspension

INTERVENTIONS:
Drug: Sisunatovir — Single Dose
  Arms: Treatment A; Treatment B
Drug: Rabeprazole 40 mg — Tablets once daily for 7 days
  Arms: Treatment B; Treatment E
Drug: Sisunatovir suspension — Tablets once daily for 7 days
  Arms: Treatment C; Treatment D; Treatment E
Drug: Rabeprazole 20 mg — Tablets once daily for 7 days
  Arms: Treatment D

SUMMARY:
The purpose of this study is to see how rabeprazole affects the level of the study medicine sisunatovir in the blood of healthy adult participants. Rabeprazole is a medicine that reduces the amount of acid the stomach makes.

The information from this study may inform how sisunatovir will be used in the future with medicines that reduce stomach acid.

This study is seeking healthy participants who:

* are aged 18 years of age or older.
* are confirmed to be healthy by some medical tests. This study can include both men and women. Women who can produce a baby must agree to use a highly effective method of birth control.
* have body mass index (BMI) of 16 to 32 kilograms per meter squared.
* a total body weight of more than 45 kilograms. Participants will receive sisunatovir tablets by mouth on Day 1. After at least 48 hours, participants will take rabeprazole tablets by mouth once a day for 7 days. On the last (7th) day of rabeprazole dosing, another dose of sisunatovir tablets will be taken by mouth.

The study will look at the blood levels of sisunatovir with and without taking rabeprazole. This will help see how sisunatovir should be given in the future.

The total planned time of participation is about 10 to 11 weeks. The study consists of:

* screening period of up to 28 days before taking sisunatovir.
* 13 days of staying in the study clinic.
* a follow-up contact that will occur 28 to 35 days after taking sisunatovir the last time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and standard 12-lead electrocardiogram (ECG).
* Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine,pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* A positive urine drug test at screening or admission.
* A positive serum pregnancy test at screening and/or positive urine/serum pregnancy test in woman/women of childbearing potential (WOCBP) at Day -1
* Current use of any prohibited concomitant medication(s) for sisunatovir and/or medication(s) that are contraindicated in the rabeprazole prescribing information.
* Use of tobacco/nicotine containing products
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest.
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR) (units of mL/min/1.73m²) <60 mL/min(/1.73m²) based on 2021 chronic kidney disease epidemiology (CKD-EPI).
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (Bili) ≥ 1.05 × upper limit of normal (ULN). Participants with an elevated total bilirubin consistent with Gilbert's Disease should have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0 to 72 hour postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | 0 to 72 hours postdose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 to 72 hours postdose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention
Number of Participants With Clinical Laboratory Abnormalities | Baseline to Study Day 12 (Part 1) or Study Day 20 (Part 2)
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline to Study Day 12 (Part 1) or Study Day 20 (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241017